CLINICAL TRIAL: NCT02072681
Title: Mild and Rapidly Improving Stroke Study
Acronym: MaRISS
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: American Heart Association (Other); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Jose Romano, MD, Professor of Clinical Neurology, University of Miami
Other Study IDs: 20120079
Record Dates: First submitted 2014-01-09; First posted 2014-02-26 (Estimated); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mild and Rapidly Improving Ischemic Stroke: Patients 18 years or older with mild or rapidly improving acute ischemic stroke defined clinically. .Absence of non-ischemic conditions neuro-imaging (i.e. absence of hemorrhage or a mass on brain imaging that arrived to the hospital within 4.5 hours after the onset of stroke symptoms.
  All participants will have two follow up telephone calls: One at approximately 30 days after the stroke and one at approximately 90 days after the stroke to ask questions about how well participant can carry out usual duties after the stroke, how much assistance do he/she needs to perform your daily activities and how good or bad would he/she considers current health to be.

SUMMARY:
The objective of this study is to determine the 90-day outcomes of mild and rapidly improving ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Mild or spontaneously rapidly improving ischemic stroke confirmed by neuroimaging
* Arrival to hospital within 4.5 hours of symptom onset
* Willing to provide consent
* Available for a telephone interview at 30 and 90 days

Exclusion Criteria:

* Onset >4.5 hours
* Unable to provide informed consent (patient or legally appointed representative
* Premorbid modified Rankin Scale >1
* Unavailable by telephone for follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic stroke defined clinically as mild and/or spontaneously rapidly improving and confirmed by neuroimaging not to have a hemorrhagic stroke with symptom onset within 4.5 hours.
Sampling Method: Non-Probability Sample
Enrollment: 2175 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients not independent at 90 days | 90 days
  The primary outcome measure is proportion of patients with a modified Rankin Scale of 2-6 at 90 days

SECONDARY OUTCOMES:
Proportion of patients with dependence or disability in activities of daily living at 90 days | 90 days
  Proportion of patients not independent in activities of daily living defined as a Barthel Index score <95
Symptomatic intracranial hemorrhage due to Alteplase | 36 hours
  Amongst those that receive intravenous Alteplase, a secondary safety measure is the proportion of patients that develop neurologic worsening development of symptomatic intracerebral hemorrhage, defined as neurological deterioration that, in the judgment of the investigator, is related to intracranial hemorrhage confirmed by CT or MRI, within 36 hours of administration of Alteplase.
Proportion of patients not independent at 30 days | 30 days
  Proportion of patients with modified Rankin Scale 2-6 at 30 days.
Quality of life by the EuroQOL EQ-5D | 90 days
  EuroQOL will be treated as a continuous measure
Stroke disability by the Stroke-Impact Scale-16 | 90 days
  SIS-16 will be treated as a continuous measure
Independence with Activities of Daily Living by the Barthel Index | 90 days
  BI will be treated as a continuous measure; pre specified analysis include proportion of patients with Barthel Index <95

CONTACTS AND LOCATIONS:
Overall Officials: Jose G Romano, MD, Principal Investigator — University of Miami
Locations (97):
- United States (97):
  - Chandler Regional Medical Center, Chandler, Arizona
  - HonorHealth, Scottsdale, Arizona
  - Long Beach Memorial Medical Center, Long Beach, California
  - Good Samaritan Hospital, Los Angeles, California
  - Kaiser Permanente South California, Los Angeles, California
  - Providence Holy Cross Medical Center, Mission Hills, California
  - Riverside University Health System Medical Center, Moreno Valley, California
  - Southern California Permanente Medical Group / Downey, Pasadena, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Kaiser Permanente Northern California (Sacramento), Sacramento, California
  - Orange County Global Medical Center, Santa Ana, California
  - Memorial Hospital Central, Colorado Springs, Colorado
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Shands Hospital- University of Florida, Gainesville, Florida
  - Osceola Regional Medical Center, Kissimmee, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Morton Plant Mease Healthcare, Tampa, Florida
  - Medical Center, Navicent Health, Macon, Georgia
  - WellStar Health System-Kennestone Hospital, Marietta, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - Alexian Brothers, Arlington Heights, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Central DuPage Hospital Association, Winfield, Illinois
  - Lutheran Hospital, Fort Wayne, Indiana
  - Parkview Research Center, Fort Wayne, Indiana
  - Methodist Hospitals, Gary, Indiana
  - St. Vincent Hospital Indianapolis, Indianapolis, Indiana
  - Wesley Medical Center, Wichita, Kansas
  - King's Daughters Medical Center, Ashland, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Norton HealthCare, Louisville, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Boston Medical Center, Boston, Massachusetts
  - Berkshire Medical Center, Pittsfield, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Ascencion-St. John Providence, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Ascension-Borgess, Kalamazoo, Michigan
  - Mississippi Baptist Medical Center, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - St. Luke's Neuroscience Institute, Kansas City, Missouri
  - Cox Medical Centers, Springfield, Missouri
  - SSM Health Care St. Louis, St Louis, Missouri
  - St. Anthony's Medical Center, St Louis, Missouri
  - Mercy Hospital St. Louis, St Louis, Missouri
  - Ocean Medical Center, Brick, New Jersey
  - Hackensack Meridian Health/Jersey Shore University Medical Center, Neptune City, New Jersey
  - St. Joseph's Regional Medical Center, Paterson, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Saint Peter's Hospital, Albany, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Mercy Hospital of Buffalo, Buffalo, New York
  - Rochester General Hospital, Rochester, New York
  - Univ of Rochester - Strong Memorial Hospital, Rochester, New York
  - Crouse Hospital, Syracuse, New York
  - Albert Einstein College of Medicine-Montefiore Medical Center, The Bronx, New York
  - Faxton St. Luke's Healthcare, Utica, New York
  - Carolinas HealthCare System, Charlotte, North Carolina
  - Carolina Healthcare Blue Ridge, Morganton, North Carolina
  - Novant Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - Mercy Hospital, Oklahoma City, Oklahoma
  - Saint Francis Hospital, Tulsa, Oklahoma
  - Kaiser Permanente Northwest Sunnyside Medical Center, Clackamas, Oregon
  - Providence St. Vincent, Portland, Oregon
  - Legacy Emanuel Medical Center, Portland, Oregon
  - UPMC Altoona, Altoona, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - UPMC Hamot, Erie, Pennsylvania
  - Pennsylvania State University / The Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Conemaugh Memorial Medical Center, Johnstown, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Seton Medical Center-Brackenridge, Austin, Texas
  - Seton Medical Center, Austin, Texas
  - St. David's Medical Center/Neuro Texas Institute, Austin, Texas
  - JPS Health Network, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Clear Lake Regional Medical Center, Webster, Texas
  - Intermountain Medical Center Neuroscience Institute, Murray, Utah
  - University of Vermont, Burlington, Vermont
  - Bon Secours Hampton Roads, Norfolk, Virginia
  - Overlake Hospital Medical Center, Bellevue, Washington
  - West Virginia University, Morgantown, West Virginia
  - Aurora BayCare Medical Center, Milwaukee, Wisconsin
  - Aurora Medical Center Grafton, Milwaukee, Wisconsin
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Romano JG, Gardener H, Campo-Bustillo I, Khan Y, Riley N, Tai S, Sacco RL, Khatri P, Smith EE, Schwamm LH. The Mild and Rapidly Improving Stroke Study (MaRISS): Rationale and design. Int J Stroke. 2019 Dec;14(9):983-986. doi: 10.1177/1747493019873595. Epub 2019 Sep 7. PMID 31496438
- [Background] Romano JG, Smith EE, Liang L, Gardener H, Camp S, Shuey L, Cook A, Campo-Bustillo I, Khatri P, Bhatt DL, Fonarow GC, Sacco RL, Schwamm LH. Outcomes in mild acute ischemic stroke treated with intravenous thrombolysis: a retrospective analysis of the Get With the Guidelines-Stroke registry. JAMA Neurol. 2015 Apr;72(4):423-31. doi: 10.1001/jamaneurol.2014.4354. PMID 25642650
- [Background] Romano JG, Smith EE, Liang L, Gardener H, Campo-Bustillo I, Khatri P, Bhatt DL, Fonarow GC, Sacco RL, Schwamm LH. Distinct Short-Term Outcomes in Patients With Mild Versus Rapidly Improving Stroke Not Treated With Thrombolytics. Stroke. 2016 May;47(5):1278-85. doi: 10.1161/STROKEAHA.115.011528. Epub 2016 Mar 17. PMID 26987870
- [Result] Romano JG, Gardener H, Campo-Bustillo I, Khan Y, Tai S, Riley N, Smith EE, Sacco RL, Khatri P, Alger HM, Mac Grory B, Gulati D, Sangha NS, Craig JM, Olds KE, Benesch CG, Kelly AG, Brehaut SS, Kansara AC, Schwamm LH; MaRISS Investigators*. Predictors of Outcomes in Patients With Mild Ischemic Stroke Symptoms: MaRISS. Stroke. 2021 Jun;52(6):1995-2004. doi: 10.1161/STROKEAHA.120.032809. Epub 2021 May 5. PMID 33947209
- [Derived] Gardener H, Romano LA, Smith EE, Campo-Bustillo I, Khan Y, Tai S, Riley N, Sacco RL, Khatri P, Alger HM, Mac Grory B, Gulati D, Sangha NS, Olds KE, Benesch CG, Kelly AG, Brehaut SS, Kansara AC, Schwamm LH, Romano JG. Functional status at 30 and 90 days after mild ischaemic stroke. Stroke Vasc Neurol. 2022 Apr 26;7(5):375-80. doi: 10.1136/svn-2021-001333. Online ahead of print. PMID 35474180
- [Derived] Romano JG, Gardener H, Smith EE, Campo-Bustillo I, Khan Y, Tai S, Riley N, Sacco RL, Khatri P, Alger HM, Mac Grory B, Gulati D, Sangha NS, Olds KE, Benesch CG, Kelly AG, Brehaut SS, Kansara AC, Schwamm LH; MaRISS Investigators*. Frequency and Prognostic Significance of Clinical Fluctuations Before Hospital Arrival in Stroke. Stroke. 2022 Feb;53(2):482-487. doi: 10.1161/STROKEAHA.121.034124. Epub 2021 Oct 14. PMID 34645285